CLINICAL TRIAL: NCT05129098
Title: Left Bundle Branch Pacing Versus Conventional Pacing in Patients With Atrioventricular Node Disorders: a Randomized, Control Study
Brief Title: Left Bundle Branch Pacing Versus Conventional Pacing in Atrioventricular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Georgios Leventopoulos, Principa Investigator, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 251/10-05-21
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Atrioventricular Nodal Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Bundle Branch Pacing (Experimental): Implantation of a left bundle branch lead via sheath, to perform left bundle branch pacing
  Interventions: Device: Left bundle branch pacing lead (Select Secure 3830 lead)
- Conventional Right Venticular Pacing (Active Comparator): The ventricular lead will be implanted in the right ventricle in the conventional way
  Interventions: Device: Right ventricular active fixation lead

INTERVENTIONS:
Device: Left bundle branch pacing lead (Select Secure 3830 lead) — Implantation of a left bundle branch pacing lead via sheath
  Arms: Left Bundle Branch Pacing
Device: Right ventricular active fixation lead — Active fixation lead (standard)
  Arms: Conventional Right Venticular Pacing

SUMMARY:
Recently, the concept of physiological pacing has emerged in the clinical practice, in an attempt to prevent the deteriorating effects of right ventricular pacing in the long-term. Left bundle branch pacing seems to be a safe procedure with promising results that may prevent intraventricular dyssynchony compared with the conventional right ventricular pacing.

DETAILED DESCRIPTION:
In this prospective, randomized study the outcomes regarding echocardiographic indices of dyssynchrony in left bundle branch versus conventional right ventricular pacing in patients with atrioventricular node disease will be compared In recent years, His pacing has demonstrated better results regarding resynchronization compared to conventional biventricular pacing in trials of 3D mapping. However, technical difficulties that relate to unstable lead positioning or inability in succeeding low pacing threshold have led to low success rates. An alternative site of physiological pacing that could possibly overcome these issues, while maintaining ventricular synchrony is left bundle branch pacing. The lead implantation of LBB pacing is performed using the Select Secure (3830) pacing lead. The lead is screwed into the interventricular septum, until left bundle branch pacing is achieved. The randomized patients 24 hours after the procedure are echocardiographically evaluated and indices of mechanical dyssynchrony are recorded. Follow-up is conducted at 3 months, 6 months and one year post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Patients with atrioventricular block and EF>50% with a predicted ventricular pacing rate>20%
* Patients with intraventricular septal diameter>8mm
* Written informed consent

Exclusion Criteria:

* Indication for CRT or ICD device
* Patients with no subclavian approach, who are candidates for leadless devices
* Presence of severe tricuspid regurgitation
* Patients who are candidates for implantation from the right side, as currently the provided tools for left bundle branch pacing fascilitate only left sided pacemaker implantations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Echocardiographic dyssynchrony index, as expressed with Global Left Ventricular Myocardial Work Efficiency (GWE) (%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the global left ventricular work efficiency- as a measure of dyssynchrony- will be recorded.

SECONDARY OUTCOMES:
Procedure Time (min) | 1 Day of procedure
  The total time required for the completion of the procedure
Fluoroscopy Time (min) | 1 Day of procedure
  The total time of fluoroscopy
Dose Area Product (DAP) (cGy/cm2) | 1 Day of procedure
  Total Radiation Dose as expressed with DAP
Implant success | 1 Day of procedure
  Successful implantation with pacing threshold<2 V
Complications associated with pacemaker implantation | through study completion at 1 year post randomisation
  General device related complications: pneumothorax, hemothorax, infection, tamponade, hematoma, lead reoperation Specific complications associated with the left bundle branch pacing procedure: intraventricular septum rupture, septal perforator branch injury with subsequent myocardial infarction or lead displacement
B natriuretic peptide measurement (pg/ml) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Blood samples are extracted in all patients at baseline, 3 months, 6 months and one year after the procedure
Stroke volume index (SVi) (ml/m2) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the SVi will be recorded
Ejection Fraction (EF) (%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the EF will be recorded
Global Longitudinal Strain (GLS) (%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the GLS will be recorded
Left Atrium Strain (%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the Left Atrium Strain will be recorded
Left Atrium Strain Rate (1/s) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the Left Atrium Strain Rate will be recorded
Aortic Time- Velocity Integral (TVI) (cm) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and the aortic TVI will be recorded
Global Work Index (GWI) (mmHg%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and GWI will be recorded
Global Constructive Work (GCW) (mmHg%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and GCW will be recorded
Global Wasted Work (GWW) (mmHg%) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and GWW will be recorded
Segmental CW, WW at the mid septal wall | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and segmental WI, CW, WW at the mid septal wall will be recorded
Segmental CW, WW at the basal lateral wall | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and segmental WI, CW, WW at the basal lateral wall will be recorded
Peak Strain Dispersion (PSD) (msec) | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  Follow-up transthoracic echocardiography will be held 24 hours, 3 months, 6 months and one year after the procedure and PSD will be recorded
Changes in capture threshold (V) in the ventricular lead | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  The device will be interrogated at baseline, 3 months, 6 months and one year after the procedure and the potential changes in capture threshold in the ventricular lead will be recorded
Changes in sense (mV) in the ventricular lead | 24 hours after the procedure as baseline and change at 3 months, 6 months and one year post-procedure
  The device will be interrogated at baseline, 3 months, 6 months and one year after the procedure and potential changes in sense in the ventricular lead will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Leventopoulos, MD, PhD, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Rion, Greece